CLINICAL TRIAL: NCT05943015
Title: Comparison of Postoperative Analgesic Efficacy of Quadratus Lumborum II, Quadratus Lumborum III and Paravertebral Blocks in Elective Laparoscopic Cholecystectomies
Brief Title: Analgesic Efficacy of Quadratus Lumborum, Paravertebral Blocks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GaziosmanpasaTREHEK
Record Dates: First submitted 2023-06-21; First posted 2023-07-12 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2024-07

CONDITIONS: Postoperative Pain
Keywords: paravertebral block; quadratus lumborum block; laparoscopic cholecystectomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Quadratus Lumborum Block II (Active Comparator): Quadratus Lumborum Block II
  Interventions: Procedure: Quadratus Lumborum Block II; Drug: Patient controlled intravenous analgesia
- Quadratus Lumborum Block III (Active Comparator): Quadratus Lumborum Block III
  Interventions: Procedure: Quadratus Lumborum Block III; Drug: Patient controlled intravenous analgesia
- Paravertebral Block (Active Comparator): Paravertebral Block
  Interventions: Procedure: Paravertebral Block; Drug: Patient controlled intravenous analgesia

INTERVENTIONS:
Procedure: Quadratus Lumborum Block II — Patients are placed in the lateral decubitus position. The area where the block will be applied is disinfected with povidine iodine. A convex ultrasound probe is placed on the midaxillary line above the iliac crest. By visualizing the psoas major and the transverse process adjacent to the quadratus lumborum muscle, using the in-plane technique, using a 22 gauge 80 mm peripheral block needle negative aspiration into the middle layer of the thoracolumbar fascia posterior to the quadratus lumborum muscle, then 0.5-1 ml of saline 20 ml of 0.25% bupivacaine will be injected after hydrodissection is observed. The same will be done to the other side.
  Arms: Quadratus Lumborum Block II
Drug: Patient controlled intravenous analgesia — Afterward of the operation, patients will be treated with patient-controlled analgesia with intravenous tramadol, with 20 mg bolus 20 minutes lock time, 4-hour limit 100 mg and 24-hour limit 400 mg
  Arms: Quadratus Lumborum Block II
Procedure: Quadratus Lumborum Block III — Patients are placed in the lateral decubitus position. The area where the block will be applied is disinfected with povidine iodine. A convex ultrasound probe is placed on the midaxillary line above the iliac crest. By visualizing the transverse process adjacent to the psoas major and quadratus lumborum muscles, using the in-plane technique, using a 22 gauge 80 mm peripheral block needle after negative aspiration into the anterior layer of the thoracolumbar fascia anterior to the quadratus lumborum muscle muscle, 0.5-1 ml of serum After observing hydrodissection with physiological, 20 ml of 0.25% bupivacaine is injected. The same is done to the opposite side.
  Arms: Quadratus Lumborum Block III
Drug: Patient controlled intravenous analgesia — Afterward of the operation, patients will be treated with patient-controlled analgesia with intravenous tramadol, with 20 mg bolus 20 minutes lock time, 4-hour limit 100 mg and 24-hour limit 400 mg
  Arms: Quadratus Lumborum Block III
Procedure: Paravertebral Block — Patients are placed in the lateral decubitus position. The area where the block will be applied is disinfected with povidine iodine. The linear ultrasound probe is placed longitudinally at the T6 level, 2-2.5 cm lateral to the spinous processes. Transverse process, superior costotransverse ligament and pleura are visualized, 22 gauge 80 mm peripheral block needle is passed with in-plane technique, superior costotransverse ligament is passed, negative aspiration into the paravertebral space under the ligament, followed by 0.5-1 ml of saline and hydrodissection of the pleura, followed by 20 ml of 0.25% bupivacaine is injected.The same is done to the opposite side.
  Arms: Paravertebral Block
Drug: Patient controlled intravenous analgesia — Afterward of the operation, patients will be treated with patient-controlled analgesia with intravenous tramadol, with 20 mg bolus 20 minutes lock time, 4-hour limit 100 mg and 24-hour limit 400 mg
  Arms: Paravertebral Block

SUMMARY:
This trial is a prospective, randomized, single-center, single blinded-analysis trial, the objective of which is compare the postoperative analgesia efficacy of Quadratus lumborum II, Quadratus Lumborum III and Paravertebral blocks in elective laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Laparoscopic approach in cholecystectomy surgery is frequently preferred because of its advantages in systemic complications, morbidity, mortality and hospital stay. Pain is one of the important causes of late discharge after surgery. Laparoscopic cholecystectomy surgery requires a multimodal analgesia approach because of its multiple pain components.Regional analgesia techniques are effective in reducing the side effects such as intraoperative opioid use, postoperative pain and nausea and vomiting. Quadratus lumborum block and paravertebral plane blocks are regional techniques performed for multimodal analgesia.

The aim of this study is to determine an effective analgesia method by comparing the postoperative analgesic effectiveness of Quadratus Lumborum II, Quadratus Lumborum III and Paravertebral blocks in elective laparoscopic cholecystectomy surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years, American Society of Anesthesiologists physical statusⅠ-II

Exclusion Criteria:

* local anesthetic allergy
* Infection at the procedure site
* Body Mass Index >35 kg/m2
* Anticoagulant use with bleeding disorder
* Chronic analgesia and opioid use
* with mental and psychiatric disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Total amount of tramadol use | within 24 hours after the surgery
  The total tramadol use of the patients in 24 hours will be recorded.

SECONDARY OUTCOMES:
Visual Analogue Scale values at 1st, 6th, 12th and 24th hours | at 1st, 6th, 12th and 24th hours after the surgery
  Visual Analogue Scale is a scale of 0-10 cm in length, expressed by non-standard verbal descriptors (no pain-unbearable pain..) indicating the limits of pain intensity on both sides, horizontally or vertically.
Block onset time | 30 min after the block
  In order to evaluate sensory block, dermatome involvement will be evaluated with ice between Thoracic 1 and Lumbar 5 levels. When the feeling of coldness disappears, dermatome involvement will be considered. The sensory block formation time with ice will be evaluated as the block onset time, the10th, 20th and 30th minute dermatome area involvement will be recorded.
intraoperative remifentanil consumption | during operation procedure
  The total remifentanil use to be used in the maintenance of 0.05-0.2 mcg/kg remifentanil will be recorded by titration according to the hemodynamic data of the intraoperative patients.
postoperative length of hospital stay | within 1 weeks after the surgery
  time to patient's discharge
side effects such as nausea, vomiting and shoulder pain | within 24 hours after the surgery
  The incidence of postoperative side effects such as nausea, vomiting and shoulder pain will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: EMINE KOSE, Principal Investigator — Gaziosmanpasa Research and Education Hospital; DONDU GENC MORALAR, Principal Investigator — Gaziosmanpasa Research and Education Hospital; SERPIL SAHIN SEHIRLIOGLU, Principal Investigator — Gaziosmanpasa Research and Education Hospital
Locations (1):
- Gaziosmanpasa Resarch and Education Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang J, Cui X, Ren L, Li X, Zhang Y, Xie Y, Ji Z, Huang Y. Comparison of the Postoperative Analgesic Effects between Ultrasound-Guided Transmuscular Quadratus Lumborum Block and Thoracic Paravertebral Block in Laparoscopic Partial Nephrectomy Patients: A Randomized, Controlled, and Noninferiority Study. Pain Res Manag. 2023 Feb 20;2023:8652596. doi: 10.1155/2023/8652596. eCollection 2023. PMID 36891030